CLINICAL TRIAL: NCT01091350
Title: Influence of Equilibration Rate Constant (ke0) of Propofol on the Effect-site Concentration for Loss of Consciousness
Brief Title: Influence of Equilibration Rate Constant (ke0) of Propofol on the Effect Site Concentration for Loss of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Hwang, MD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Orchestra vs Diprifusor
Record Dates: First submitted 2010-03-14; First posted 2010-03-24 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Diprifusor group (Active Comparator): Propofol was infused via Diprifusor TCI (Target-controlled infusion)
  Interventions: Device: Diprifusor (Target-controlled infusion)
- Orchestra group (Experimental): Propofol was infused via Orchestra TCI
  Interventions: Device: Orchestra (Target-controlled infusion)

INTERVENTIONS:
Device: Diprifusor (Target-controlled infusion) — Two TCI devices with different Teo and same Marsh PK model
  Other Names: Diprifusor(Grasby Medical Limited, United Kingdom)
  Arms: Diprifusor group
Device: Orchestra (Target-controlled infusion) — Two TCI devices with different Teo and same Marsh PK model
  Other Names: OrchestraTM (Fresenius Vial, Brezins, France)
  Arms: Orchestra group

SUMMARY:
The aim of this study is to validate that an effect compartment concentration for loss of consciousness (LOC) was varied according to different Keo value.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing general anesthesia

Exclusion Criteria:

* Hepatic or renal disease
* Drug addiction

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Estimated effect-site propofol concentration at loss of consciousness | after propofol infusion

SECONDARY OUTCOMES:
Time to loss of consciousness | after propofol infusion